CLINICAL TRIAL: NCT00990392
Title: Pilot Study: Topical Antibiotics for Prevention of ICU Central Line Infections
Brief Title: Topical Antibiotics for Prevention of Intensive Care Unit (ICU) Central Line Infections
Acronym: ToPICL
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Change of practice to antibiotic impregnated catheters and large study published showing their efficacy. Made topical antibiotics obselete.
Sponsor: Fraser Health (Other)
Responsible Party: Principal Investigator, Steve Reynolds, Critical care Physician, Fraser Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Kerrie-333333
Record Dates: First submitted 2009-10-05; First posted 2009-10-06 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Blood Stream Infections; Skin Diseases, Infectious
Keywords: Blood stream infections; Catheter related infections; Central venous catheter related infections; Line sepsis; Topical antibiotics; Bacitracin; Polymixin; Gramicidin; Polysporin Triple Therapy; Intensive care unit
MeSH Terms: conditions — Skin Diseases, Infectious; Catheter-Related Infections | interventions — Gramicidin; Bacitracin; Petrolatum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Polysporin Triple Therapy (Experimental): Polysporin Triple Therapy ointment applied to the insertion point at the time of CVC placement and twice within the first week.
  Interventions: Drug: Polysporin Triple Therapy ointment
- Placebo (Placebo Comparator): Petroleum jelly
  Interventions: Other: Petroleum Jelly

INTERVENTIONS:
Drug: Polysporin Triple Therapy ointment — Polysporin Triple Therapy ointment applied to the insertion point at the time of CVC placement and twice within the first week.
  Other Names: Polysporin Triple Therapy (gramicidin, polymixin, bacitracin)
  Arms: Polysporin Triple Therapy
Other: Petroleum Jelly — Petroleum jelly applied to the insertion point at the time of CVC placement and twice within the first week.
  Other Names: Vaseline
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine if the overall central venous catheter related infection rate can be reduced by the application of Polysporin Triple Therapy ointment to the insertion site.

DETAILED DESCRIPTION:
Previous studies in the dialysis population have found a reduction in local and system central venous catheter related infections with the application of topical antibiotics to the insertion point. One such study found a mortality benefit with Polysporin Triple Therapy ointment. We intend to determine if this preparation can reduce overall line infection rates in the ICU environment through its application at the time of line insertion and twice more the following week.

ELIGIBILITY:
Inclusion Criteria:

* all patients admitted to the ICU requiring a central venous catheter

Exclusion Criteria:

* previous line infection during same ICU stay
* CVC for hemodialysis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-11; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Overall number of line related infections (local and blood borne) | 6 months

SECONDARY OUTCOMES:
Length of ICU stay | 7 months
Length of hospital stay | 7 months
Prevalence of methicillin-resistant Staphylococcus Aureus (MRSA) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Steven Reynolds, MD, Principal Investigator — Fraser Health Authority
Locations (1):
- Royal Columbian Hospital, New Westminster, British Columbia, Canada

REFERENCES:
- [Background] Lok CE, Stanley KE, Hux JE, Richardson R, Tobe SW, Conly J. Hemodialysis infection prevention with polysporin ointment. J Am Soc Nephrol. 2003 Jan;14(1):169-79. doi: 10.1097/01.asn.0000038688.76195.a4. PMID 12506149
- [Background] James MT, Conley J, Tonelli M, Manns BJ, MacRae J, Hemmelgarn BR; Alberta Kidney Disease Network. Meta-analysis: antibiotics for prophylaxis against hemodialysis catheter-related infections. Ann Intern Med. 2008 Apr 15;148(8):596-605. doi: 10.7326/0003-4819-148-8-200804150-00004. PMID 18413621